CLINICAL TRIAL: NCT01323166
Title: Retrospective Study of APR Results Regarding Patients' Self Reported Quality of Life
Brief Title: Quality of Life After Abdominoperineal Resection for Rectal Cancer, Comparing Two Surgical Techniques
Acronym: APR
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Swedish Cancer Foundation (Other)
Responsible Party: Principal Investigator, Eva Angenete, M.D., Ph.D., Sahlgrenska University Hospital
Other Study IDs: QoL after APR at SU
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Rectal Cancer
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Excision of the levator muscle: The abdominal part of the operation is performed as an TME and the perineal part of the operation is performed with the intent to get a cylindrical specimen thus removing part of or the entire levator muscle with the specimen
  Interventions: Procedure: Excision of the levator muscle
- Traditional perineal operation: The abdominal part of the operation performed as a TME. The perineal operation performed with the intent of removing the tumour with CRM free of tumour and the levator left in place
  Interventions: Procedure: Excision of the levator muscle

INTERVENTIONS:
Procedure: Excision of the levator muscle — Cylindrical perineal excision including the levator muscle
  Other Names: Abdomino perineal resection; Extra levator excision; Perineal excision

SUMMARY:
The purpose of the study is to compare self-reported health related quality of life after two different operating techniques for low rectal cancer operated by rectal amputation, using a specific and detailed questionnaire. The population has been operated over a 6 year period in one university hospital.

DETAILED DESCRIPTION:
Low rectal cancer treated by abdominoperineal resection (APR, rectal amputation)has worse prognosis than other rectal cancers, both regarding local recurrence and cancer specific survival. With a view to improve local recurrence rates a more extensive perineal operation (excision of the levator muscle) has been suggested. In our university hospital thie technique was introduced for all surgeons January 2007. A population of all patients operated from 1 January 2007 to 31 December 2009 was compared to all patients operated from 1 January 2004 to 31 December 2006 using the traditional, less extensive method, in all a six year period and 158 patients.

A specific questionnaire was developed after in depth interviews, and was face-validated by patients who had undergone an APR. This questionnaire will be sent out to all patients in our population who are still alive.

The patients will be contacted first by a letter of invitation, later called by telephone to be given more information and asked for permission to send the questionnaire.

The send out of invitation letters will start March 2011.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer operated by abdominoperineal resection 2004-2009

Exclusion Criteria:

* no informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: colorectal section of one university hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of life after rectal cancer surgery - possible differences due to choice of procedure | 2-7 years after operation
  A detailed questionnaire with 250 questions, where emphasis is on physical satisfaction and emotional status as well as bowel function, sexual function and stoma function 2-7 years after rectal amputation

SECONDARY OUTCOMES:
Impact of rectal cancer surgery on household finances in a long-term perspective | 2-7 years after operation
  Part of the questionnaire deals with the patients'/spouses' career and economic situation after the operation.
Impact of rectal cancer surgery and the level of intrusive thoughts | 2-7 years after operation
  Part of the questionnaire analyses occurrence and effects of intsrusice thoughts

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, MD,PhD, Principal Investigator — Dept. of Surgery, Sahlgernska Univesity Hospital/Ostra
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

REFERENCES:
- [Derived] Angenete E, Asplund D, Andersson J, Haglind E. Self reported experience of sexual function and quality after abdominoperineal excision in a prospective cohort. Int J Surg. 2014 Nov;12(11):1221-7. doi: 10.1016/j.ijsu.2014.10.003. Epub 2014 Oct 12. PMID 25311774